CLINICAL TRIAL: NCT05097404
Title: Clinical Utility of Vesical Imaging Report and Data System (VI-RADS) in Diagnosis of Muscle Invasive Bladder Cancer
Brief Title: Clinical Utility of VI-RADS in Diagnosis of MIBC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SamsungMC_UroRadiology
Record Dates: First submitted 2021-09-27; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-09

CONDITIONS: Radical Cystectomy; Muscle-Invasive Bladder Carcinoma; Multiparametric MRI; Vesical Imaging Report and Data System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bladder Cancer (BCa) is the 9th most common cancer worldwide. In general, BCa is presented as a non-muscle invasive bladder cancer (NMIBC) in 70% of patients and treated with transurethral resection of bladder tumor (TUR-BT). However, in cases of muscle invasive bladder cancer (MIBC), radical cystectomy (RC) is the gold standard of treatment. Therefore, It is important to distinguish MIBC from NMIBC.

To date, pathologic staging is based on the result of TUR-BT before RC. However, it is operator dependent, thus residual cancer may be remained depending on surgical experience. Therefore, about 7%-30% patients of MIBC can be underestimated with NMIBC, and it can be increased to 45% if the muscle is not resected. Consequently, it has been raised the need for imaging test to overcome diagnostic limitations.

Multiparametric magnetic resonance imaging (mpMRI) has been widely used in the field of diagnosis of BCa. In 2018, the Vesical Imaging Report and Data System (VI-RADS) was published using T2-weighted imaging (T2WI), diffusion-weighted imaging (DWI), and dynamic contrast enhanced (DCE) imaging, and 5-point VI-RADS scoring system has been proposed and reported as an imaging test useful for assessing muscle involvement in primary bladder cancer Therefore, in this study, we investigate the diagnostic performance of the VI-RADS scoring system that can differentiate NMIBC from MIBC in primary bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* primary bladder cancer in cystoscopy
* suitable for MRI and TUR-BT
* agreement to participate in the study and signing of an informed consent form

Exclusion Criteria:

* history of TUR-BT
* previous radiation and/or chemotherapy for bladder cancer
* Not suitable for MRI or TUR-BT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary bladder cancer Healthy suitable to perform multiparametric MRI pre-operatively Perform TUR-BT that has been sufficiently implemented to check for muscle invasion
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of VI-RADS scoring system in diagnosis of MIBC | From Sep 2021 to Sep 2024
  diagnostic accuracy of VI-RADS scoring system in diagnosis of MIBC

SECONDARY OUTCOMES:
clinical utility of VI-RADS to predict adverse pathology after repeat TUR-BT in high risk NMIBC | From Sep 2021 to Sep 2024
  clinical utility of VI-RADS to predict MIBC after repeat TUR-BT in high risk NMIBC (To predict the chance of MIBC after repeat TUR-BC according to VI-RADS score in patients with high risk MNIBC)
clinical utility of VI-RADS to reduce unnecessary repeat TUR-BT in high risk NMIBC | From Sep 2021 to Sep 2024
  clinical utility of VI-RADS to reduce unnecessary repeat TUR-BT in high risk NMIBC (To predict the chance of NMIBC after repeat TUR-BC according to VI-RADS score in patients with high risk MNIBC)
Prediction of MIBC according to the VI-RADS scoring system | From Sep 2021 to Sep 2024
  Prediction of MIBC according to the VI-RADS scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Antoni S, Ferlay J, Soerjomataram I, Znaor A, Jemal A, Bray F. Bladder Cancer Incidence and Mortality: A Global Overview and Recent Trends. Eur Urol. 2017 Jan;71(1):96-108. doi: 10.1016/j.eururo.2016.06.010. Epub 2016 Jun 28. PMID 27370177
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Divrik RT, Sahin AF, Yildirim U, Altok M, Zorlu F. Impact of routine second transurethral resection on the long-term outcome of patients with newly diagnosed pT1 urothelial carcinoma with respect to recurrence, progression rate, and disease-specific survival: a prospective randomised clinical trial. Eur Urol. 2010 Aug;58(2):185-90. doi: 10.1016/j.eururo.2010.03.007. Epub 2010 Mar 19. PMID 20303646
- [Background] Shindo T, Masumori N, Kitamura H, Tanaka T, Fukuta F, Hasegawa T, Yanase M, Miyake M, Miyao N, Takahashi A, Matsukawa M, Taguchi K, Shigyo M, Kunishima Y, Tachiki H, Tsukamoto T. Clinical significance of definite muscle layer in TUR specimen for evaluating progression rate in T1G3 bladder cancer: multicenter retrospective study by the Sapporo Medical University Urologic Oncology Consortium (SUOC). World J Urol. 2014 Oct;32(5):1281-5. doi: 10.1007/s00345-013-1205-1. Epub 2013 Nov 5. PMID 24190368
- [Background] Panebianco V, Narumi Y, Altun E, Bochner BH, Efstathiou JA, Hafeez S, Huddart R, Kennish S, Lerner S, Montironi R, Muglia VF, Salomon G, Thomas S, Vargas HA, Witjes JA, Takeuchi M, Barentsz J, Catto JWF. Multiparametric Magnetic Resonance Imaging for Bladder Cancer: Development of VI-RADS (Vesical Imaging-Reporting And Data System). Eur Urol. 2018 Sep;74(3):294-306. doi: 10.1016/j.eururo.2018.04.029. Epub 2018 May 10. PMID 29755006
- [Background] Pecoraro M, Takeuchi M, Vargas HA, Muglia VF, Cipollari S, Catalano C, Panebianco V. Overview of VI-RADS in Bladder Cancer. AJR Am J Roentgenol. 2020 Jun;214(6):1259-1268. doi: 10.2214/AJR.20.22763. Epub 2020 Apr 14. PMID 32286874
- [Background] Del Giudice F, Barchetti G, De Berardinis E, Pecoraro M, Salvo V, Simone G, Sciarra A, Leonardo C, Gallucci M, Catalano C, Catto JWF, Panebianco V. Prospective Assessment of Vesical Imaging Reporting and Data System (VI-RADS) and Its Clinical Impact on the Management of High-risk Non-muscle-invasive Bladder Cancer Patients Candidate for Repeated Transurethral Resection. Eur Urol. 2020 Jan;77(1):101-109. doi: 10.1016/j.eururo.2019.09.029. Epub 2019 Nov 5. PMID 31699526